CLINICAL TRIAL: NCT05769374
Title: Effects of Parental Involvement in Active Video Games Play on Physical Activity, Psychosocial Beliefs and Parent-child Relational Quality on Overweight and Obese Male Adolescents in China
Brief Title: Effects of Parental Involvement in Exergames Play on Physical and Mental Health on Overweight and Obese Male Adolescent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Mai Yiqiang, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Mai Yiqiang
Record Dates: First submitted 2023-02-18; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Physical Inactivity; Overweight and Obesity; Psychosocial Problem
Keywords: Parental involvement; Exergame; Physical activity; Psychosocial
MeSH Terms: conditions — Sedentary Behavior; Overweight; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: In this experiment, experiment group 1 is AVG with parents' participation, that is, the experiment object is accompanied by parents to complete the experiment, and experiment group 2 is to complete the experiment task by themselves under the supervision of parents. The control group did not undergo any AVG intervention and maintained the same physical activity as usual.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Two player mode(parental involvement) in AVG play (Experimental): the parent involvement group requires one parent to accompany the child to complete the experimental task
  Interventions: Device: cooperative versus competitive AVG play
- Single player mode in AVG play (Experimental): the single-person model and the child need to complete the experimental task under the parent's supervision.
  Interventions: Device: cooperative versus competitive AVG play
- children did not engage in any AVGs play (Active Comparator): children did not engage in any AVGs play nor any other structured school-based PA programs beyond physical education.
  Interventions: Device: cooperative versus competitive AVG play

INTERVENTIONS:
Device: cooperative versus competitive AVG play — The duration of the study was 8 weeks and the frequency was 60 minutes three times a week. In the first two weeks, three games, Golf, Just Dance and Tennis, will be selected to experiment on easy and normal difficulty respectively. In the three weeks from week 3 to Week 5, Bowling, Shape Boxing and Table tennis will be selected for the experiment with easy, normal and difficult difficulties respectively. In the last three weeks, Rowing, Family ski and Baseball will be selected to carry out experiments with easy, ordinary and difficult difficulty respectively.Additionally,participants in control group did not participate in any AVG intervention and maintained their daily physical activity behaviors

SUMMARY:
In recent years, with the rising obesity rate, overweight and obesity have become a hot issue of public health. As a sensitive and special group, teenagers shoulder the heavy responsibility of building the motherland, so their health is also the focus of scholars and experts. As a new type of sports game, active video game(AVG) has been proved by many studies to be able to effectively improve the sedentary behavior of teenagers, and can completely become a substitute for today's popular smart phones. In addition, due to the increase of overweight and obese teenagers, a series of psychological problems, such as anxiety, depression, and low self-esteem, also troubled this group. Some researchers can effectively improve the psychological status of the subjects through the intervention experiment of AVG. However, there are few studies on psychosocial beliefs at present, and the impact of psychosocial variables such as self-efficacy, social support and quality of life on overweight and obese groups is extremely important. Moreover, due to the impact of the COVID-19 epidemic, the relationship between family members will also change, especially the alienation and rigidity of the relationship between children and parents will show a significant growth trend. Therefore, this study mainly takes AVG play with parents' participation as the main intervention means to influence the physical activities, psychosocial beliefs and quality of parent-child relationship of the experimental target.

DETAILED DESCRIPTION:
In this study, three groups, namely the control group (children did not engage in any AVGs play nor any other structured school-based PA programs beyond physical education), two experimental groups (parental involvement in AVG play and single-player mode). It should be noted that the parent involvement group requires one parent to accompany the child to complete the experimental task, while the single-person model and the child need to complete the experimental task under the parent's supervision. The sample is 13-14-year-old Chinese overweight and obese male middle school students. Researchers will establish three groups in the WeChat platform to facilitate communication with each group of experimental subjects.

A study of 73 previously inactive, typically developing children showed initially high intrinsic motivation to use an AVGs system, which disappeared by week seven of the survey. However, the overall results of a study indicate that the use of AVGs may have increased self-reported levels of PA in overweight or obese children over 12 weeks. Given that the group in this study is junior high school students in grade one or two, with heavy learning tasks, the research period is eight weeks.

Based on the articles, according to the characteristics of the Nintendo Wii, to increase the subject's compliance with the game and maximize the training effect, each gaming session consisted of the upper body, cardio,and sports games . Routines were pre-determined and varied daily, gradually increasing in difficulty throughout the program. AVG participants were tracked every time for individual progress in the two experimental groups by earning points and expending calories, which were continuously reported by the Wii console as the participants played. After each game session, the parents will export the data from the game console and send it to the researcher through WeChat.

ELIGIBILITY:
Inclusion Criteria:

* The family needs to install a television and connect to the Internet
* The family has never purchased a game console similar to AVG before
* ensure that at least one parent has enough time to accompany his or her child to complete the experimental task in a week
* BMI percentile should be more than 85
* there are no other sports besides daily physical activities
* The parents of the subjects agreed with their children to participate in the experiment and were willing to participate with their children.

Exclusion Criteria:

* Clinically diagnosed with mental illness
* Clinically diagnosed chronic disease
* Relevant weight loss drugs taken within half a year

Ages: 13 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-04-10 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Questionnaire for Children (PAQ-C) | Before the experiment
  It is a self-filled and retrospective physical activity level questionnaire for children and adolescents (PAQ-C)(aged 7 to 18). On the one hand, PAQ-C measures the general level of physical activity by scoring (continuous variable) rather than measuring the intensity, frequency, and duration of physical activity, which improves its operational and theoretical feasibility; On the other hand, PAQ-C helps to improve time efficiency and reduce capital costs, making it easy to manage and operate.Likert's 5-level scoring method adopted five numbers of scores from 1(strongly disagree) to 5 (strongly agree) were used, and the scores were converted into linear scales. Higher scores indicated the higher PA level.
Pediatric Quality of Life Inventory 4.0 (PedsQL) | Before the experiment
  The scale is used to assess the quality of life of young adults in the past seven days. The scale included 23 items, which assessed the physical (8 items), social (5 items), school (5 items), and emotional (5 items). Likert's 5-level scoring method adopted five numbers of scores from 0 (never) to 4 (almost always) were used, and the scores were converted into linear scales. Higher scores indicated the higher quality of life.
The Self-Efficacy for School Physical Activity Questionnaire | Before the experiment
  Physical activity efficacy scale [the Self-Efficacy for School Physical Activity Questionnaire (SEPAQ)] to assess task related efficacy in the main school activity behavioural.Using the scale, please check the appropriate response (0-100%) for each question.Higher scores indicated the higher self-efficacy level
Parent child relational quality scale | Before the experiment
  From the perspective of adolescents, this scale includes 29 items and is divided into four dimensions: parent-child intimacy, parent-child conflict, parent-child trust, and parent-child satisfaction to measure the quality of the parent-child relationship.
  Scoring: This questionnaire adopts a 5-point Likert scale, with 1-5 representing increasing support (1=strongly disagree; 2=Disagree;3=Not necessarily;4=agree; 5=strongly agree).Higher scores indicated the higher parent child relational quality
Parental Support Scale for Children's Physical Exercise | Before the experiment
  The questionnaire includes 20 items. From the parent's perspective, parents' support for children's physical activity behavior is measured from five dimensions: verbal encouragement, physical activity model, logistical support, behavior encouragement, and physical activity preference.
  Scoring: This questionnaire adopts a 5-point Likert scale, with 1-5 representing increasing support (1=never; 2=rarely; 3=sometimes; 4=often; 5=always.Higher scores indicated the higher parental support level

SECONDARY OUTCOMES:
Physical Activity Questionnaire for Children (PAQ-C) | Mid-test:end of week 4
  It is a self-filled and retrospective physical activity level questionnaire for children and adolescents (PAQ-C)(aged 7 to 18). On the one hand, PAQ-C measures the general level of physical activity by scoring (continuous variable) rather than measuring the intensity, frequency, and duration of physical activity, which improves its operational and theoretical feasibility; On the other hand, PAQ-C helps to improve time efficiency and reduce capital costs, making it easy to manage and operate.Likert's 5-level scoring method adopted five numbers of scores from 1(strongly disagree) to 5 (strongly agree) were used, and the scores were converted into linear scales. Higher scores indicated the higher PA level.
Pediatric Quality of Life Inventory 4.0 (PedsQL) | Mid-test:end of week 4
  The scale is used to assess the quality of life of young adults in the past seven days. The scale included 23 items, which assessed the physical (8 items), social (5 items), school (5 items), and emotional (5 items). Likert's 5-level scoring method adopted five numbers of scores from 0 (never) to 4 (almost always) were used, and the scores were converted into linear scales. Higher scores indicated the higher quality of life.
The Self-Efficacy for School Physical Activity Questionnaire | Mid-test:end of week 4
  Physical activity efficacy scale [the Self-Efficacy for School Physical Activity Questionnaire (SEPAQ)] to assess task related efficacy in the main school activity behavioural.Using the scale, please check the appropriate response (0-100%) for each question.Higher scores indicated the higher self-efficacy level
Parent child relational quality scale | Mid-test:end of week 4
  From the perspective of adolescents, this scale includes 29 items and is divided into four dimensions: parent-child intimacy, parent-child conflict, parent-child trust, and parent-child satisfaction to measure the quality of the parent-child relationship.
  Scoring: This questionnaire adopts a 5-point Likert scale, with 1-5 representing increasing support (1=strongly disagree; 2=Disagree;3=Not necessarily;4=agree; 5=strongly agree).Higher scores indicated the higher parent child relational quality
Parental Support Scale for Children's Physical Exercise | Mid-test:end of week 4
  The questionnaire includes 20 items. From the parent's perspective, parents' support for children's physical activity behavior is measured from five dimensions: verbal encouragement, physical activity model, logistical support, behavior encouragement, and physical activity preference.
  Scoring: This questionnaire adopts a 5-point Likert scale, with 1-5 representing increasing support (1=never; 2=rarely; 3=sometimes; 4=often; 5=always.Higher scores indicated the higher parental support level

OTHER OUTCOMES:
Physical Activity Questionnaire for Children (PAQ-C) | Post-test:end of week 8
  It is a self-filled and retrospective physical activity level questionnaire for children and adolescents (PAQ-C)(aged 7 to 18). On the one hand, PAQ-C measures the general level of physical activity by scoring (continuous variable) rather than measuring the intensity, frequency, and duration of physical activity, which improves its operational and theoretical feasibility; On the other hand, PAQ-C helps to improve time efficiency and reduce capital costs, making it easy to manage and operate.Likert's 5-level scoring method adopted five numbers of scores from 1(strongly disagree) to 5 (strongly agree) were used, and the scores were converted into linear scales. Higher scores indicated the higher PA level.
Pediatric Quality of Life Inventory 4.0 (PedsQL) | Post-test:end of week 8
  The scale is used to assess the quality of life of young adults in the past seven days. The scale included 23 items, which assessed the physical (8 items), social (5 items), school (5 items), and emotional (5 items). Likert's 5-level scoring method adopted five numbers of scores from 0 (never) to 4 (almost always) were used, and the scores were converted into linear scales. Higher scores indicated the higher quality of life.
The Self-Efficacy for School Physical Activity Questionnaire | Post-test:end of week 8
  Physical activity efficacy scale [the Self-Efficacy for School Physical Activity Questionnaire (SEPAQ)] to assess task related efficacy in the main school activity behavioural.Using the scale, please check the appropriate response (0-100%) for each question.Higher scores indicated the higher self-efficacy level
Parent child relational quality scale | Post-test:end of week 8
  From the perspective of adolescents, this scale includes 29 items and is divided into four dimensions: parent-child intimacy, parent-child conflict, parent-child trust, and parent-child satisfaction to measure the quality of the parent-child relationship.
  Scoring: This questionnaire adopts a 5-point Likert scale, with 1-5 representing increasing support (1=strongly disagree; 2=Disagree;3=Not necessarily;4=agree; 5=strongly agree).Higher scores indicated the higher parent child relational quality
Parental Support Scale for Children's Physical Exercise | Post-test:end of week 8
  The questionnaire includes 20 items. From the parent's perspective, parents' support for children's physical activity behavior is measured from five dimensions: verbal encouragement, physical activity model, logistical support, behavior encouragement, and physical activity preference.
  Scoring: This questionnaire adopts a 5-point Likert scale, with 1-5 representing increasing support (1=never; 2=rarely; 3=sometimes; 4=often; 5=always.Higher scores indicated the higher parental support level

CONTACTS AND LOCATIONS:
Overall Officials: Yiqiang Mai, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Universiti Putra Malaysia, Jiaozuo, Henan, China

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I don't want to share it until after graduation

REFERENCES:
- [Result] Takeuchi H, Taki Y, Hashizume H, Asano K, Asano M, Sassa Y, Yokota S, Kotozaki Y, Nouchi R, Kawashima R. The impact of television viewing on brain structures: cross-sectional and longitudinal analyses. Cereb Cortex. 2015 May;25(5):1188-97. doi: 10.1093/cercor/bht315. Epub 2013 Nov 20. PMID 24256892
- [Result] Staiano AE, Marker AM, Beyl RA, Hsia DS, Katzmarzyk PT, Newton RL. A randomized controlled trial of dance exergaming for exercise training in overweight and obese adolescent girls. Pediatr Obes. 2017 Apr;12(2):120-128. doi: 10.1111/ijpo.12117. Epub 2016 Feb 26. PMID 26918815
- [Result] Staiano AE, Beyl RA, Hsia DS, Katzmarzyk PT, Newton RL Jr. A 12-week randomized controlled pilot study of dance exergaming in a group: Influence on psychosocial factors in adolescent girls. Cyberpsychology (Brno). 2018;12(2):3. doi: 10.5817/CP2018-2-3. PMID 31367239